CLINICAL TRIAL: NCT01627652
Title: Human Adaptation to High Altitude
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zurich Center for Integrative Human Physiology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EK 2011-N-51
Record Dates: First submitted 2012-05-04; First posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Hypoxia
Keywords: hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Altitude

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- altitude (Experimental): subjects will be studies at sea level and at high altitude
  Interventions: Other: altitude

INTERVENTIONS:
Other: altitude — the subjects will live one month at 3450 m altitude in the Jungfraujoch Research Station
  Other Names: Jungfraujoch Research Station

SUMMARY:
This scientific study aims at studying human adaptations to high altitude and the studies will be conducted at the University of Zürich and during a 4 week high altitude "expedition" to the Jungfraujoch research station at 3450 m altitude. The proposal is made up of several independent biological research projects to be conducted in the same healthy volunteers participating in the study. Thus, the subjects will be studied at sea level, and then during 4 weeks of acclimatization to high altitude, and for some experimental purposes all subjects will also be studied one and two weeks after return to sea level.

DETAILED DESCRIPTION:
Study aim A: Red cell mass and hypoxia:

Various forms of altitude training have been used to increase in particular endurance performance of elite athletes. The most commonly used approaches is either to live and train at altitude (Live high - train high; LHTH) or to live at high altitude while training at sea level (Live high - train low; LHTL). While it is generally accepted that the potential performance enhancing effects of LHTH and LHTL are mediated through a hypoxia dependent increase in red cell mass (1), this has never been demonstrated experimentally. In 2010 the investigators conducted the first placebo controlled double blinded LHTL study (supported with BASPO funding) with the clear aim to identify the mechanism(s) responsible for the performance enchantment following LHTL. In brief, for this reason 16 elite athletes (average VO2max ≈ 70 ml.kg.min) resided for 16 hours/day in either normoxia or at the stimulated altitude of 3000 m for four weeks. This protocol was chosen based on recent reviews by experts within the field (2). Despite this supposedly optimal setting the investigators did not find a single positive change induced by LHTL. To our big surprise and despite having measured VO2max, time trial performance, red cell mass, markers of erythropoiesis at a much higher frequency than in any other previous LHTL study they all remained unaffected by LHTL. Based on our experience within altitude physiology and studies including erythropoietin injections in humans, the investigators have begun to speculate if even 3 weeks of continuous altitude exposure is sufficient stimulus to increases red cell mass which is the cornerstone assumption for LHTL (1, 3). If this is not the case, then the scientific rationale to perform LHTL vanishes.

The initial determination of red cell mass at altitude dates 100 years back when Douglas (4) reported that 6 weeks of exposure to 2300 m altitude on the Gran Canaries did not increase red cell mass whereas htc did increase. Some 50 years later Lawrence (5) concluded that a true increase in red cell mass required several weeks (8) of altitude exposure (3800 m), whereas the decrease in plasma volume begins upon arrival. It should here be noted that they used a superb method to determine red cell mass: autologous red cells tagged with radioactive phosphorous, something that is not possible today. In 1964 Hannon (6) conducted his now classic study when he exposed 8 female and 8 males to 4300 m altitude for 9 full weeks. During the first month there was no increase in red cell mass, and over the next 5 weeks red cell mass only increased by 5% despite of continued iron supplementation. The method used in this particular study was autologous chromium-51-labbeled red cells, i.e. gold standard. Even at the severely high altitude of 5450 m (with no relevance for elite sport), Reynafarje (7) reported that 6 weeks are required for an increase in red cell volume. To follow up on all previous altitude studies is impossible here, but in a recent review Grover and Bärtsch (8) summarized these by stating that "True polycythemia develops when residence at high altitude (3800-4500m) extends over months to years". Thus, as compared to the altitude research done in the past in regards to red cell mass, mostly conducted with the use of techniques by far superior to those used today and at higher latitudes than applied in LHTL protocols, the proposal that LHTL should increase red cell mass seems at odds. It should be kept in mind however, that in most altitude studies it is difficult to isolate the effects to hypoxia, and also changes in temperature, nutritional intake and physical activity level are often a confounding factor.

Levine and Stray-Gundersen (3) were the first to report an increase in red cell mass following LHTL. After 3 weeks of LHTL at 2500 m they calculated RCV to be increased by 8% based on changes in plasma volume as derived by Evens Blue. Evens blue is a poor measure for changes in RCV since it rapidly leaks from the circulation, and the data should be taken with some caution. It is also interesting that an increase in RCV was only observed in 50% of the LHTL subjects. This does not exclude that the observed changes were simply not just the result of biological variation (9). In the 10 years following the first positive LHTL results the data could not be replicated. Especially the Australian research group lead by Chris Gore made huge efforts in this period but could not confirm that 3 weeks of LHTH or normobaric LHTL caused RCV to increase (10-16). From 2006 and onwards positive effects of LHTL have been reported on RCV, but the data are far from convincing. The research group of J.P. Richalet conducted a series of experiments in Premanon, and found red cell mass to increase in one study (17), but unchanged in another two studies (18, 19). J Wehrlin from the Bundesamt für Sport found three weeks of LHTL to increase RCV (20), but the study design is not clean as subjects from different disciplines served as control and treatment subjects. This is a problem since they were at different stages in their training season and it cannot be excluded that this does not affect RCV. Since the subjects were elite athletes competing at the international level it is also a pity that no anti-doping samples were collected in this subject's population. Chris Gore has for the last few years applied an unusual statistical approach and thereby reported what they call "marginal" increases in RCV following LHTL (21). This conclusion however cannot be drawn if using a standard accepted statistical approach. Thus, although it is generally accepted that LHTL may increase RCV, the picture is not as clear as expected, and the investigators argue that it is rather unlikely when comparing with the above mentioned chronic altitude exposure studies.

The main aim with this present study is to determine in a large study population (n=16) if continuous exposure to 3450 m altitude for four weeks increases red cell mass or not. The investigators have chosen this altitude because 1) In populations living permanently at this altitude, an elevated red cell volume has been reported as compared to their countrymen living near sea level, 2) If the investigators choose a lower altitude, and the investigators observe no increase in red cell mass the investigators would not be able to determine whether this was the consequence of a too low altitude or a too short exposure duration, 3) Exposure to much higher elevations may not be suitable for athletes.

Study protocol for Study aim A: Red cell mass and hypoxia One month before altitude exposure subjects will on a weekly basis have their RCV (by CO rebreathing) and other hematological parameters quantified on two separate days not separated by more than one day (i.e. Monday and Tuesday, or Tuesday and Wednesday etc). This allows for a very good estimation of their basal hematological values. Light iron supplementation (40 mg/day will be started on day 1 and kept throughout the study). Furthermore, all subjects will perform light bike exercise at 1.0 W/kg body weight for 30 minutes every second day during this month. Such light activity is known not to influence red cell mass (22). The activity will be continued during the altitude exposure period at the Jungfraujoch (see below), in order to limit any potential effect altitude/confinement induced physical inactivity which may induce a decrease in plasma volume, which however is reported to be eliminated by even very light (23). On two occasions/week while at Jungfraujoch all subjects will be escorted to the Mönchhütte (same altitude) and back (total 60 min of walking) in order to also keep some physical activity. While at altitude all subjects will perform the same test as at sea level, i.e. double determination of hematological parameters on a weekly basis.

Study aim B: Cardiovascular adjustments to high altitude:

Classic studies by Grollman on Pikes Peak ( 4300m) in the US demonstrated that there is an approximately 40% increase in resting cardiac output (heart rate × stroke volume) within the first days of ascent to high altitude (Grollman 1930). Similar observations have been made under more rigorously controlled conditions in the laboratory, with equivalent degrees of hypoxia (24, 25). Changes in stroke volume play a minor role in the altitude induced increase in cardiac output, and most of the response (90-95%) seems to be the result of an increase heart rate (24, 25). Following a few days of altitude exposure however, cardiac output returns to sea level values or to even lower values despite hypoxemia is still persisting (26). The decrease in cardiac output is surprising and occurs despite an continuous increased heart rate and is a consequence of a reduction in stroke volume (26, 27). Similar data are reported with exercise, i.e. a decrease in stroke volume with submaximal and maximal exercise (28). The physiological mechanism leading to a reduction in stroke volume at rest and during exercise with continuous exposure to high altitude remains unknown, and the main aim with Study B is to resolve this issue. Since cardiac output to a large degree depends on blood volume (Frank-Starling mechanism) and left ventricular filling, it is tempting to speculate that the altitude dependent decrease in plasma volume and hence also total blood volume causes right ventricle filling and subsequently also stroke volume to be reduced. To test this hypothesis to interventions will be performed:

1. To facilitate venous return, and hence right ventricle filling, subjects will on a weekly basis be tested on the commonly used tilt-table. The tilt table allows investigation of subjects in the supine position at various head-down tilts. The investigators wish to study our volunteers during 5 minutes of head down tilt at (at each tilt) -15, -30 and -45°, which is normal procedure. The head down tilt facilitates venous return and hence stroke volume. The largest effects are usually seen at around -70°. During the last minute of each tilt cardiac output will be assess by an inert re-breathing technique (the investigators have had this procedure approved by the ETH ethical board in previous applications) and by ultra sound doppler. Heart rate and blood pressure will continuously be monitored non-invasively.
2. On the last study day at the Jungfraujoch plasma volume will be restored to sea level values by infusion of Dextran. The exact volume of dextran to be infused is calculated by multiplying the red cell volumes (assessed in project A) with the hematocrit. Cardiac output will be assessed as above in the supine and seated position before and immediately after the infusion of Dextran.
3. Stroke volume and heart rate will be determined during submaximal and maximal exercise by inert-gas re-breathing on a weekly basis during acclimatization. The investigators hypothesize that the expected changes in stroke volume correlate well with altitude induced changes in plasma and blood volume.

Study C: Autonomic nervous control at high altitude:

Exposure to hypoxia causes sympathoexcitation in humans. This has been determined indirectly by measurements of the hypoxia-induced increases in noradrenaline (Cunningham et al., 1965) and directly by increases in muscle sympathetic nerve activity (Saito et al., 1988). The primary underlying mechanism is activation of chemoreceptors in the carotid body (Marshall, 1994) and the brainstem (Solomon, 2000). Thus, during acute exposure to hypoxia, heart rate and sympathetic nerve activity change significantly when blood oxygen saturation decrease to about 85% (Smith et al., 1996). In humans, this level of saturation results from breathing hypoxic gas mixtures with an FIO2 of 0.11-0.13 with some individual variation (Lundby et al., 2004). Recently it was demonstrated that sea level residents acclimatizing for 4 weeks to an altitude of 5260m above sea level exhibited a surprisingly high level of muscle sympathetic nerve activity (Hansen & Sander, 2003). The average muscle sympathetic burst frequency increased to 300% above sea level values, which is considerably more than the 50-100% expected during acute exposure to a corresponding hypoxic gas mixture (FIO2 0.105). One limitation to this first study was the inclusion of only one time-point during the altitude acclimatization. Thus, it is unknown whether high altitude sympathoexcitation as measured by microneurography subsides during further acclimatization in sea level residents.

The specific mechanisms underlying this apparent high altitude sympathoexcitation are unclear. Concurrent breathing of pure oxygen and intravenous infusion of saline at high altitude to restore blood homeostasis only caused a minor decrease in muscle sympathetic nerve activity (Hansen & Sander, 2003), suggesting that traditional activation of the peripheral chemoreflex or the cardiopulmonary baroreflex do not account for the sympathoexcitation. In stead, chronic exposure to hypoxia may cause resetting of the central nervous pathways involved in sympathoexcitatory reflexes. There is a growing body of evidence supporting that pharmacologically-induced inhibition of brainstem nitric oxide signalling causes amplification or resetting of sympathoexcitatory reflexes, and it has been suggested that accumulation of endogenous inhibitors of nitric oxide could be similarly involved in human sympathoexcitatory states.

The underlying mechanism of high altitude sympathoexcitation (point 1-5 below)

It is unknown how chronic hypoxia causes sympathoexcitation, but some of the potential underlying mechanisms are described below:

1. Arterial baroreflex-activation. In previous high altitude MSNA-studies the sea level residents had minor but significant increases in arterial blood pressure of about 8-12mmHg (29, 30), which rules out arterial baroreflex unloading. Resetting of the arterial baroreflex has not been ruled out as a contributing factor, but it is unlikely as a major mechanism.
2. Cardiopulmonary baroreflex-activation. In a chronic high altitude study (29), an intravenous infusion of saline (800-1000ml over 15 min) caused only a small decrease in sympathetic traffic, providing evidence that unloading of cardiopulmonary baroreceptors is not a primary contributor.
3. Chemoreflex-sensitization. The ventilatory and sympathoexcitatory responses to high altitude acclimatization share several characteristics. Both responses develop gradually over days, and once established normalization is slow over days after re-exposure to normoxia (29, 31, 32). Ventilatory and sympathetic chemoreflexes share the afferent input from peripheral chemoreceptors, and the central neuronal circuitries responsible for efferent activation of phrenic nerves and sympathetic outflow are parallel. The investigators hypothesize that hyperventilatory and sympathoexcitatory responses to chronic hypoxic exposure share underlying mechanisms. Ventilatory acclimatization to high altitude is thought to primarilly depend on chemoreflex-sensitization, i.e. despite stable or even slightly improving arterial oxygen tension during the first 2 weeks of acclimatization, the hypoxic chemoreflex ventilatory response (HVR) slowly is augmented. The basis for this unique reflex-sensitization has been studied quite extensively over the last several decades. In humans, it is likely that both peripheral and central mechanisms are involved.

   Peripherally, the signaling events in the chemoreceptors within carotid and aortic bodies are complex involving several excitatory and inhibitory transmitters. The excitatory signals include adenosine, ATP, acetylcholine and endothelin. The primary inhibitory signaling molecules are dopamine (acting on D2-receptors, D2R) (33), noradrenaline, and NO. In humans, intravenous low-dose dopamine and the D2R-antagonist domperidone (now only administered orally) are able to decrease and augment sea level HVR, respectively (34, 35), but not maximal hypoxic ventilation (36). Neither low-dose dopamine or domperidone cross the blood-brain barrier. Although, dopamine production and effects within the carotid body may decrease during the first days of hypoxic exposure (37, 38), enzymes involved in dopamine production, dopamine receptors, and dopamine-concentration (and noradrenaline) are upregulated during chronic hypoxia (38). The functional consequence for ventilatory responses in humans have been studied sparingly, but one study suggests that the effects of both dopamine and dompridone on HVR are unaltered or slightly larger in subjects exposed to hypoxia for 8h (35). The role of NO in peripheral chemoreception has not been studied in humans, but recent animals studies suggest the peripheral inhibitory action of NO is confounded by NO-mediated disinhibition of dopamine-effects. Thus, sodium nitroprusside actually increase peripheral chemoreceptor firing in cats perhaps by blocking endogenous dopamine-inhibition (39).

   Centrally, chemoreceptor-afferent activation causes release of L-glutamate and dopamine within the nucleus tractus solitarii (NTS). These events lead to excitation of NTS-neurons that in turn via L-glutamate excite brainstem neurons within the rostral ventrolateral medulla (RVLM). The collected input to RVLM-neurons control the central sympathetic outflow from the brainstem. Animal studies have suggested that modulation of the chemoreflex pathway within NTS by dopamine (excitatory) (40) nitric oxide (NO) (excitatory) (41) becomes more significant during hypoxic exposure. Thus microinjection of sodium nitroprusside and the NO synthase inhibitor L-NMMA into NTS in awake rats cause an increase and a decrease in ventilation during hypoxic exposure (41). The role of central D2R in hypoxia have been studied in rats by comparing HVR after domperidone (peripheral D2R blockade) with HVR after domperidone + haloperidol (a peripheral and centrally acting D2R blocker) (42). The overall effects of haloperidol alone on the ventilatory response to isocapnic hypoxia in humans was a reduction in HVR (43).

   While a number of neuronal pathways and transmitters both peripherally and centrally may play physiological roles in chemoreflex-sensitization linked to altitude-acclimatization, recent studies in D2R-knock-out mice have provided compelling evidence that D2R are a prerequisite (44). For this reason the present study will test whether sensitization of the chemoreceptors is an underlying cause for high altitude sympathoexcitation, and if so whether dopamine- or NO-related mechanisms are involved. In this regard, it should be noted that, acute hyperoxia or even three days of normoxic breathing failed to normalize sympathetic traffic in healthy subjects acclimatized to high altitude for 4 weeks (29). However, similar findings have been reported for ventilation. Thus, chronic hypoxia may cause such a substantial sensitization of the chemoreflex, that even hyperoxia may fail to silence the primary peripheral chemoafferents from the carotid and aortic bodies, and it has been speculated that hyperoxia may actually cause central excitation of ventilatory and sympathetic output after acclimatization to altitude.
4. Decreased NO-production in brainstem-vasomotor centers. Soon after it was discovered that NO was an important endothelium-derived vasodilator, NO also emerged as a neuromodulator augmenting glutamatergic neurotransmission (45). It has since been well established in animal models that the overall functional significance of NO deficiency within brain stem centers is sympathoexcitation and augmentation of sympathoexcitatory reflexes (46). This form of sympathoexcitation has been identified in humans (47). Thus, while some studies indicate an increased NO-production within NTS, the overall NO-production could be decreased during hypoxic exposure. Indeed, a recent human study have suggested that there is at least a relative NO-deficiency with lower blood cGMP-levels during hypoxic exposure (48). In a high altitude study, intravenous infusion of the NO substrate, L-arginine, had no effect on sympathetic traffic (Lundby et al., 2002abstract). This finding does not exclude NO-deficiency during chronic hypoxia, but merely indicates that such putative deficiency is not related to a relative lack of the substrate for NO synthesis. The present study adresses this unresolved issue in two independent ways. First, whole-body NO-production will be determined by a novel stable-isotope technique. Second, L-NAME will be is used to produce NO synthase inhibition. Under ambient air conditions this will reveal whether the functional significance of endogenous NO-production is decreased in chronic hypoxia. During HVR-testing L-NAME may have complex effects on the chemoreflex due to both disinhibition at the level of the peripheral chemoreceptors and indirect inhibitory action within NTS of the brainstem.
5. Neurophysiological characteristics of high altitude sympathoexcitation The high altitude sympathoexcitation has not yet been characterised using single-unit recordings. The single-unit characteristics such as firing probability and probabilities of dual and multiple single-unit firing within one heart cycle will allow cross-sectional comparison of sympathetic traffic between lowlanders and high altitude natives. Furthermore, sympathetic single-unit characteristics have recently been published for the sympathoexcitatory states of heart failure, sleep apnoea, and hypertension (49). Thus, important comparisons can be made to other sympathoexcitatory states. The firing characteristics may have important implications for noradrenaline release.

Peripheral uncoupling of sympathetic activity and vasomotor tone Despite a dramatic increase in sympathetic nerve activity, and noradrenaline release, there is a limited (albeit statistically significant) increase in vascular resistance and blood pressure at high altitude. This is logically related to hypoxia-induced peripheral offsetting of sympathetic vasoconstriction. The uncoupling could be caused at least partially by alpha-receptor downregulation, although there was no significant decrease in cardiac alpha-1-receptors in rats living in hypobaric hypoxia for 21 days (50). In addition, acute severe hypoxic exposure also causes an uncoupling of sympathetic activity and vasomotor tone. Thus, in humans using FiO2 of 0.08, sympathetic traffic is very high, but vascular resistance and blood pressure are decreased (51). This acute hypoxia effect is unlikely to be explained by receptor downregulation.

Hypotheses for high altitude sympathoexcitation tested with the proposed application:

1. The high altitude sympathoexcitation will be characterised by an increased probability of sympathetic single-unit firing, resembling characteristics of sympathoexcitation in heart failure.
2. Chronic hypoxic exposure causes substantial sensitisation of the chemoreflex, which at least partially explains the sympathoexcitation of high altitude.

3a) Central nervous D2R-mediated dopamine effects are importantly involved in chemoreflex sensitisation in high altitude sympathoexcitation.

3b) Altered NO-signaling is importantly involved in chemoreflex sensitisation in high altitude sympathoexcitation.

Hypotheses for peripheral uncoupling of sympathetic responses 4) Chronic hypoxic exposure causes decreased local and whole body nitric oxide production.

Volunteers will be each studied 4 times (2 control studies in Zürich, with and without L-NAME, and 2 studies at Jungfraujoch in week 3), with and without L-NAME.

Each study day will include the following:

Meaurements: BP, HR, Plethysmographic limb blood flow, Ventilation (incl oxygen uptake), Pulseoximetry, and MSNA single-units, and MSNA multi-units for the full chemoreflex-study. Blood samples: Including: Catecholamines, RBC-channels, cGMP.

Condition:

* Rest
* Chemoreflex (6 different oxygen levels in arterial blood) (protocol suggested by Mou et al. 1995).

NB-1: CO2 will be kept at ambient breathing levels (i.e. the resting value measured in each individual), by adding small amounts of CO2 during the chemoreflex tests.

NB-2: On one study day, intravenous dopamine-infusion (3 µg kg -1 min-1) (Dahan et al. 1996), domperidone-tablets (0,75 mg kg-1) (Pedersen et al. 1999, Lundby et al. 2001), and intravenous metoclopramide (10 mg) (Takeuchi et al. 1993) will be used in this sequence at sea level and at Jungfraujoch to inhibit and disinhibit peripheral chemoafferent firing, and subsequently inhibit central D2R-related chemoreflex excitation. Dopamine effects disappear within a few minutes after stopping infusion (Dahan et al. 1996, Jarnberg et al. 1981). Domperidone effects will reach maximum about 30 minutes after tablet ingestion, and remain fairly stable for another 30 minutes. At these doses, dopamine and domperidone do not cross the blood-brain barrier and consequently the contribution of central sensors of hypoxia is unaltered. Metoclopramide has been reported to cause an increase in sympathetic activity at sea level. If the investigators confirm this after domperidone-treatment at sea level, any decrease in sympathetic traffic in high altitude will strongly suggest hypoxia-related changes in central D2R-related chemoreflex excitation.

Study aim D: Skeletal muscle and adipose tissue metabolic adjustments to high altitude:

Hypoxia-dependent control of mitochondrial function has long been of interest however surprisingly little is known regarding this topic in either humans or animals. Previous observations of mitochondrial modifications following acclimatization to altitude (especially high and extreme altitudes) have been inconsistent. Initial reports (52-55) demonstrated greater expression of indirect markers suggestive of enhanced oxidative potential in both animals and humans native to high altitude, leading investigators to postulate that acclimatization may improve respiratory capacity and mitochondrial function in response to an increasingly hypoxic environment (55). This initial paradigm was challenged when further studies of lowlanders sojourning to high/extreme altitudes reported either a dramatic loss of skeletal muscle mitochondria (56, 57) or negligible changes in mitochondrial profile following acclimatization to high/extreme altitude (58-62), even despite significant reductions in skeletal muscle mass (60, 61). One consistency across the literature, however, has been the assumption that mitochondrial function (i.e. respiratory capacity, substrate control of respiration, and efficiency or coupling control) is represented via static measurements alone such as mitochondrial specific protein concentrations/activity or morphometric analysis representing mitochondrial content or volume, respectively. While such static measurements are not to be discounted, as they are vital to the study and our understanding of mitochondrial physiology, relying on these measurements for the characterization of mitochondrial function and oxidative potential is incomplete. Examination of mitochondrial function requires direct specific manipulations of mitochondrial respiration so potential changes in oxidative phosphorylation and electron transport can be identified. Alterations in whole body protein turnover (63) and hypoxia facilitated changes in protein concentration, including several mitochondrial proteins (64) from this study have already been reported. To elucidate hypoxia induced changes in skeletal muscle mitochondrial function following acclimatization to high altitude, the investigators wish to assess mitochondrial function of permeabilized skeletal muscle fibers and adipose tissue at sea level and after approximately 20-24 days of exposure to high altitude.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 yrs of age
* male
* healthy

Exclusion Criteria:

* smokers

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-07 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Human adaptation to high altitude | May-June, 2012
  The primary outcome measure are changes in red cell blood mass, cardiac output, middle cerebral blood flow, muscle sympathetic activity and mitochondrial function.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zürich and the JUngfraujoch Research Station, Zürich and Jungfraujoch (mountain), Switzerland